CLINICAL TRIAL: NCT00255476
Title: A Randomised Phase II Study to Investigate the Feasibility and Benefits of Combining ZD1839 and Cisplatin/5FU, as Induction Therapy, in Patients With Locally and Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: The IRESSA Novel Head and Neck Chemotherapy Evaluation Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0544
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Squamous Cell Cancer; Cancer of Head and Neck
MeSH Terms: conditions — Neoplasms, Squamous Cell; Head and Neck Neoplasms | interventions — Gefitinib; Cisplatin

INTERVENTIONS:
Drug: gefitinib
Drug: cisplatin
Drug: 5-flourouracil

SUMMARY:
The purpose of this study is to compare the objectie tumour response rate between the cisplatin/5FU and cisplatin/5FU plus ZD1839 combination

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Patients with histologically proven primary SCCHN
* Aged 18 or over

Exclusion Criteria:

* Patients eligible for surgery with curative intent
* Other co-existing malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Exclude UCNT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 2004-02; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To compare the objective tumour response rate between cisplatin/5FU and cisplatin/5FU and ZD1839 combination in these patients

SECONDARY OUTCOMES:
To compare safety and tolerability in these patients

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Iressa Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, London, United Kingdom